CLINICAL TRIAL: NCT07086482
Title: Effect of Cyanoacrylate Tissue Adhesive Versus Collagen Sponge on Palatal Donor Site Healing After Harvesting a Free Gingival Graft: a Randomized Controlled Clinical Trial
Brief Title: Effect of Cyanoacrylate Tissue Adhesive Versus Collagen Sponge on Palatal Donor Site Healing
Acronym: RCT
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Beirut Arab University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-H-0140-D-M-0588
Record Dates: First submitted 2025-07-18; First posted 2025-07-25 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Palate; Wound
Keywords: palatal donor area; Cyanoacrylate glue; wound healing; free gingival graft
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Collagen sponge (Active Comparator): Participants will be treated with collagen sponge at the palatal donor wound to achieve hemostasis. After FGG harvest, pressure will be applied at the palatal wound using a gauze soaked in saline to top the bleeding, then a collagen sponge will be placed and stabilized with 4/0 silk (x) sutures.
  Interventions: Device: Collagen sponge
- Cyanoacrylate tissue adhesive (Experimental): Participants will be treated with cyanoacrylate tissue adhesive (PeriAcryl) at the palatal donor wound to achieve hemostasis. After FGG harvest, pressure will be applied at the palatal wound using a gauze soaked in saline to top the bleeding, then PeriAcryl will be applied with a pipette following manufacturer's instructions on the entire area of the wound.
  Interventions: Combination Product: Cyanoacrylate tissue adhesive

INTERVENTIONS:
Combination Product: Cyanoacrylate tissue adhesive — Cyanoacrylate tissue adhesive is a chemical synthetic and hybrid tissue sealant possessing strong, rapid acting adhesive properties and is often used in general surgery. Recently, cyanoacrylate tissue adhesive has been effectively introduced into dentistry to close wounds and stop ischemic areas from forming in periodontal aesthetic surgeries. As well as in exposed membranes to preserve the bone graft after guided bone regeneration, in post-extraction sockets, and to seal any surgical flap. This material has strong hemostatic, bacteriostatic, and sealing qualities.
  Other Names: PeriAcryl
  Arms: Cyanoacrylate tissue adhesive
Device: Collagen sponge — Collagen sponge is an organic polymer that promotes the development of blood clots, and it resorbs quickly and completely over time. Collagen sponge create a matrix at the bleeding site, encourage platelet activation and aggregation, and engage the extrinsic coagulation pathway. Thus, it can be utilized as the first choice for wound healing.
  Arms: Collagen sponge

SUMMARY:
The goal of this clinical trial is to learn if the use of cyanoacrylate glue (PeriAcryl) is effective in healing of the palatal donor site in adults requiring a free gingival graft.

The main question[s] it aims to answer [is/are]:

Does PeriAcryl accelerate the palatal tissue healing compared with the use of collagen sponge? Does PeriAcryl usage leave the patients more satisfied?

Researcher will compare the outcomes of participants treated with PeriAcryl to those treated with collagen sponge to see if PeriAcryl accelerated the healing process of palatal tissues and led to fewer postoperative complications.

Participants will:

* be assigned to a study group using PeriAcryl or control group using Collagen sponge.
* be followed-up to monitor healing and gather clinical information.

DETAILED DESCRIPTION:
This study investigates new approaches to make management of the palatal donor area easier to the operator and more comfortable to the patient. More specifically, it compares the use of PeriAcryl glue (PA) to the use of collagen sponge after harvesting a free gingival graft from the palate in terms of wound healing and epithelization primarily, and patients satisfaction and oral health related quality of life secondarily.

Participants selection:

Healthy patients (with no systemic diseases or coagulation disorders) requiring a free gingival graft to treat a gingival recession or keratinized tissue deficiency around implants and natural teeth will be recruited.

Participants included in this study must have clinically healthy gingiva and good oral hygiene.

Participants grouping:

* Control group: Hemostasis will be achieved by collagen sponge stabilized with 4/0 silk (x) suture on the palatal wound.
* Test group: Cyanoacrylate tissue adhesive (Periacryl®, GluStitch Inc., Canada) will be applied with a pipette following manufacturer's instructions on the entire area of the wound.

All the procedures will be achieved with the full knowledge and consent of the patient. A written informed consent will be obtained for each patient included in this study.

Surgical Protocol:

* Full mouth scaling will be done for every patient at least 2 weeks before the surgery.
* The donor area will be anesthetized using articaine 4% with epinephrine 1:100,000.
* Palatal tissue thickness will be measured using a periodontal probe. Then a free gingival graft (FGG) will be harvested using a 15c blade of 1 to 1.5 mm in thickness, approximately 3 mm away from the palatal gingival margin.
* Pressure will be applied to the donor surface using gauze soaked in saline solution to stop bleeding, while the FGG will be prepared, stabilized and sutured at the recipient site.
* The operator will then receive a sealed envelope holding each patient's assigned grouping as soon as the graft extraction process is finished.

Post-operative Care:

All patients will get the same prescription of antibiotics (Amoxiclave 1g) twice daily for 7 days, and Ibuprofen 600 mg every 8 hours only taken when needed. As well as chlorohexidine 0.12% mouthwash twice daily for 2 weeks.

The same instructions will be given to all the patients (cease smoking, soft diet, oral hygiene, not brushing hard and causing trauma to the surgical site...).

The test group participants receiving PA in the palatal donor will be informed about the material and that it will disintegrate on its own after 10 days.

While the control group participants receiving collagen sponge with (x) sutures in the palatal donor will be informed that the sutures will be removed after 2 weeks.

Following the operation, a questionnaire will be given to each patient asking them to record any spontaneous bleeding of the surgical incision during the first seven days following the procedure, as well as to rate their level of postoperative discomfort using a visual analogue scale (VAS), quantity of analgesics taken, and other questions related to quality of life.

Follow-ups:

All patients will be followed-up at 7, 14, 21 days, 1 month, 2 months, and 3 months, to evaluate healing up to the formation of the first epithelial layer as evaluated by pressure with a periodontal probe and Laundry wound healing index, and the time of complete integrity of the treated palatal fibromucosa.

ELIGIBILITY:
Inclusion Criteria:

* Low-moderate anesthetic risk (ASA I-II)
* No restriction on ethnicity or gender
* Patients requiring FGG from the palate for periodontal plastic surgery
* Clinically healthy gingiva after phase I therapy
* Full-mouth plaque index grades 0 and 1
* Bleeding scores <15%

Exclusion Criteria:

* Patients who smoke > 10 cigarettes/day
* Patients with coagulation disorders
* Systemic diseases
* Patients on certain medications that may affect periodontal tissues
* Pregnant and lactating patient
* Patients with allergies to drugs that will be prescribed during the treatment phase
* Pathological mental conditions (dementia, psychosis) and lack of cooperation
* Excessive gag reflex

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
Healing of palatal wound | 1 month, 2 months and 3 months post-operatively.
  Healing will be evaluated using Laundry Wound Healing Index (WHI). WHI has a score range of 1 (very poor) to 5 (excellent), evaluates tissue color, response to palpation, presence of granulation tissue, epithelialization of incision margins, and amount of suppuration.
Epithelization of the palatal wound | On every follow-up session: 7 days, 14 days, 21 days, 1 month, 2 months and 3 months post-operatively.
  The complete epithelialization will be evaluated clinically by applying 3% hydrogen peroxide into the palatal wound. If bubble formation is not observed, epithelization will be recorded as complete, whereas if bubbles are observed, epithelization will be recorded as incomplete.
Color Match | 3 months post-operatively
  Tissue color match (CM) will be assessed with adjacent and contralateral palatal tissue (0-no color matching to 10-excellent color matching).

SECONDARY OUTCOMES:
Post-operative Pain | Every day for 7 days, and on the 14th day.
  Postoperative pain will be evaluated on a Visual analogue scale VAS (0 = no pain to 10 = worst imaginable pain).
Inflammation Degree | Every day for 7 days, and on the 14th day.
  Inflammation degree will be measured on a verbal rating scale (VRS) (0 = no inflammation, 1 = mild inflammation, 2 = marked inflammation, and 3 = extreme inflammation).
Post-operative Bleeding | Every day for 7 days, and on the 14th day.
  Spontaneous bleeding or postoperative delayed bleeding will be assessed (no: no spontaneous bleeding/yes: there is spontaneous bleeding).
Presence of Hyperesthesia | Every day for 7 days, and on the 14th day.
  Presence of hyperesthesia will be evaluated using a Verbal Rating Scale VRS (1 = none; 2 = mild, with no interference in normal life activities; and 3 = severe, with interference in normal life activities).
Number of Analgesic Pills Taken | During the first 14 days post-operatively.
  Number of analgesic pills taken by the patient post-operatively will be recorded. Minimal amount of analgesic pills taken indicate minimal post-operative pain, whereas excess use of analgesic pills indicate increased post-operative pain.
Oral Health related Quality of Life | During the first 14 days post-operatively.
  A questionnaire will be given to the participants to evaluate how the surgery affected patients' daily activities, physical state, psychological state, and oral hygiene performance. The questions will be answered with very often, fairly often, occasionally, hardly ever, never, and don't know.

CONTACTS AND LOCATIONS:
Overall Officials: Nayer Aboelsaad, Study Chair — Professor
Locations (1):
- Beirut Arab University, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Undecided